CLINICAL TRIAL: NCT04511377
Title: New Model of Short-term Rehabilitation Exercise Training Using Digital Healthcare System in Patients With Rotator Cuff Repair; Randomized Controlled Study
Brief Title: Rehabilitation Exercise Using Digital Healthcare System in Patients With Rotator Cuff Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Ministry of Health, Republic of Korea (Other Government)
Responsible Party: Principal Investigator, Jae-Young Lim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-2005/612-001
Record Dates: First submitted 2020-08-09; First posted 2020-08-13 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Rotator Cuff Tears
Keywords: Rotator Cuff Repair; Post-Operative Rehabilitation; Digital Healthcare System
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Healthcare System Rehabilitation (Experimental): Rehabilitation using Uincare Homeplus
  Interventions: Device: Rehabilitation using Digital Healthcare System (Uincare Homeplus)
- Conventional Rehabilitation (Active Comparator): Rehabilitation using Brochure
  Interventions: Other: Conventional Rehabilitation

INTERVENTIONS:
Device: Rehabilitation using Digital Healthcare System (Uincare Homeplus) — Uincare Homeplus is a device using infrared, kinect camera and motion capture technology to track 3D motion of the patients' posture and joint articulations. It also has embedded exercise training software dedicated to rotator cuff repair post-op rehabilitation at home.
  Home-based self-rehabilitation using brochure for 6 weeks post surgery (same as the active comparator)
  Home-based self-rehabilitation using digital healthcare system(Uincare Homeplus) for 6 to 12 weeks post surgery.
  Other Names: Uincare Homeplus
  Arms: Digital Healthcare System Rehabilitation
Other: Conventional Rehabilitation — Home-based self-rehabilitation using brochure for 12 weeks post surgery.
  Arms: Conventional Rehabilitation

SUMMARY:
The study aims to examine the effect of short-term rehabilitation exercise support using digital healthcare system (Uincare homeplus) in the patients with rotator cuff repair surgery. The study is a two-arm prospective randomized controlled study comparing the effect of rehabilitation exercise digital healthcare system at home with conventional brochure-based home exercise. Simple Shoulder Test (SST), Pain (using Numerical rating scale), shoulder range of motion (ROM), Disability of Arm, Shoulder and Hand (DASH), Shoulder Pain and Disability Index (SPADI), quality of life using EQ-5D will be evaluation on enrollment, 6-weeks, 12-weeks and 24-weeks after enrollment.

DETAILED DESCRIPTION:
Rotator cuff tear is one of the most common disorders affecting shoulder pain and disabilities of daily life. It is a disorder that can be caused by trauma, overuse, inappropriate usage of shoulder as well as degenerative change, which is increasing due to enlarged geriatric population. Current method of post-operative rehabilitation is home-based self rehabilitation using brochure, combined with one or two times of education at the hospital before discharge. Patients often find difficulty in doing rehabilitation by themselves at home without supervision which resulted in decreased compliance.

With development of technologies using multi-motion sensor and AR(augmented-reality) system, the investigators have developed a digital healthcare system(Uincare Homeplus) which can supplement patients' rehabilitation at home by giving them proper instructions as well as feedback.

In this prospective randomized controlled study, the investigators aimed to compare the efficacy of the newly-developed digital healthcare system with conventional rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Patient who had rotator cuff repair surgery
* Patient who is discharged to home after surgery

Exclusion Criteria:

* Patient who has previous history of shoulder surgery on the affected shoulder
* Patient who has severe neurological deficit or infection on the affected shoulder
* Patient who has severe comorbidities (Ex: uncontrolled diabetes mellitus or rheumatoid arthritis) that inhibit affected shoulder rehabilitation
* Patient who cannot participate rehabilitation program

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Estimated)
Dates: Start 2020-07-30 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Simple Shoulder Test (SST) on the affected shoulder | Enrollment, 6-weeks, 12-weeks, 24-weeks
  Simple Shoulder Test is a self-reported shoulder-specific questionnaire that measures functional limitations of the affected shoulder in patients with shoulder dysfunction. The SST consists of 12 questions with dichotomous (yes/ no) response options. score ranges from 0 to 100, higher score meaning better shoulder function.

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) on the affected shoulder | Enrollment, 6-weeks, 12-weeks, 24-weeks
  Evaluation of pain of the affected shoulder using numerical rating scale (0-10, with score 0 indicating no pain), higher scores mean worse outcome.
Range of Motion (ROM) on the affected shoulder | Enrollment, 6-weeks, 12-weeks, 24-weeks
  Evaluation of change of ROM in the affected shoulder from baseline to 24 weeks
Manual Muscle Test (MMT) on the affected arm | Enrollment, 6-weeks, 12-weeks, 24-weeks
  Evaluation of change of MMT in the affected arm from baseline to 24 weeks Upper extremities MMT ranges from 0-25, higher scoring meaning better outcome.
Disabilities of the Arm, Shoulder and Hand (DASH) on the affected arm | Enrollment, 6-weeks, 12-weeks, 24-weeks
  The DASH is a 30-item self-report questionnaire designed to assess musculoskeletal disorders of the upper limb. The score ranges from 0 (no disability) to 100 (most severe disability) with higher score meaning worse outcome.
Shoulder Pain and Disability Index (SPADI) on the affected shoulder | Enrollment, 6-weeks, 12-weeks, 24-weeks
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities.
  Overall total scores range from 0 to 130 with higher score indicating more shoulder dysfunction.
Quality of Life using EQ-5D-5L | Enrollment, 6-weeks, 12-weeks, 24-weeks
  Evaluation of quality of life using EQ-5D-5L. This scale is numbered from -0.066 to 0.904. lower value means worse quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chang WK, Lee JI, Hwang JH, Lim JY. Post-operative rehabilitation using a digital healthcare system in patients who had undergone rotator cuff repair: protocol for a single-center randomized controlled trial. Trials. 2022 Aug 17;23(1):667. doi: 10.1186/s13063-022-06648-4. PMID 35978437